CLINICAL TRIAL: NCT00275795
Title: Screening for Food Allergy, Sensitivity and Intolerances Using IgE-Specific Antigen Test and NST-NAET®
Brief Title: NAET Screening for Food Allergy, Sensitivity and Intolerances Using IgE-Specific Antigen Test and NST- NAET®
Status: Completed | Type: Observational
Sponsor: Nambudripad's Allergy Research Foundation (Other)
Other Study IDs: NAET Testing for Food Allergy; narfoundationstudy 103
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2006-11-01 (Estimated); Status verified 2006-04

CONDITIONS: Food Sensitivities; Headache; Backache; Indigestion; Eczema, Acne, Hives and Itching of the Skin
Keywords: NST-NAET testing; Food Ssensitivities; Eczema; Acne; Indigestion
MeSH Terms: conditions — Headache; Back Pain; Dyspepsia; Eczema; Acne Vulgaris; Urticaria

STUDY DESIGN:
Time Perspective: Other

INTERVENTIONS:
Procedure: NAET Procedures

SUMMARY:
Food allergy reactions cause various health disorders in sensitive people. These reactions may be IgE-mediated,cell-mediated, energy disturbance-mediated, or a combination of the three. Certain laboratory diagnostic procedures have been able to identify most IgE-mediated or cell-mediated food reactions, but so far there is no test available in traditional medicine to test the energy-mediated allergies and sensitivities. NAET® procedures have been able to identify food substances triggering to energ disturbances in sensitive people causing related health disorders. NAET uses one of the testing procedures called NST (Neuromuscular sensitivity testing).The efficacy of NST-NAET to screen food sensitivity will be evaluated in comparison with one of the well accepted, established, traditional medicine allergy testing known as the IgE-specific antigen test.

DETAILED DESCRIPTION:
Forty-two volunteers responded for an advertisement posted on the NAET web site and in the community college news bulletin board inviting them to take part in the study. They were asked to complete the NAET® Allergy Symptom-Rating (ASR) questionnaire upon arrival at the research center. Observing inclusion and exclusion criteria, a total of 32 subjects from both sexes with varied health problems were selected out of the forty-two who volunteered for the study. All 32 subjects were tested for 21 commonly used food substances via NST. Out of 32 tested, 26 subjects tested positive for one item each, from the 21 items tested and six subjects tested positive for multiple items from the selected food list. The 32 subjects had a total of 50 positive NSTs out of 672 (21X32) tests performed. The items that produced positive results by NST were further evaluated via laboratory blood serum analysis for IgE-specific antigens. According to NST the percentage of observed total food reactions in this group of 32 was 7.44%. Soon after the completion of NST the laboratory technicians collected blood from 32 subjects for IgE-specific antigen study on 50 positively tested items. The IgE-specific antigen tests were found positive on a total of 49 out of 50 tests performed.

ELIGIBILITY:
Inclusion Criteria:

A history of previous allergic reactions to one or more food substances from the selected list ( Almond, Apple, Banana, Beef, Carrot, Celery, Chocolate, Corn, Cow's milk, Crab, Egg white, Lobster, Orange, Oyster, Peanut, Salmon, Shrimp, Soybean, String bean, Tomato, and Wheat) was considered as the primary important factor for the study.

-

Exclusion Criteria:

1. Serious illnesses e.g.. Cancer, chronic obstructive pulmonary diseases, kidney diseases, heart diseases, history of anaphylaxis to any of the listed item in the inclusion criteria, mental disorders, and pregnancy.
2. Previous treatment for food allergies.
3. Knowledge of procedure -

Ages: 2 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42
Dates: Start 2005-07; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Devi S Nambudripad, DCLAcPhD, Principal Investigator — NAR Foundation
Locations (1):
- NAET Pain Clinic, Buena Park, California, United States

REFERENCES:
- [Result] Devi S. Nambudripad, M.D., Ph.D., D.C., L. Ac., Kris K. Nambudripad, BSEE, M.Ac., L.Ac, Mala M. Moosad, R.N., L.Ac., N.D., Mohan K. Moosad, DBA., M.Ac., N.D., Will Brucks, L.Ac., and Anthony DeSiena, D.C. The journal of NAET Energetics and Complementary Medicine 1(2):119-138, 2005